CLINICAL TRIAL: NCT02903316
Title: Predicting Fluid Responsiveness in on Pump Coronary Artery Bypass Graft Using Extra Systoles and Investigation of a Novel Mini Fluid Challenge Ability to Predict Fluid Responsiveness
Brief Title: Predicting Fluid Responsiveness in on Pump Coronary Artery Bypass Graft Using Extra Systoles
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 53665
Record Dates: First submitted 2016-09-05; First posted 2016-09-16 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2016-09

CONDITIONS: Hypovolemia; Coronary Artery Disease; Fluid Overload
Keywords: Fluid responsiveness; Perioperative; Extra systoles; Coronary artery bypass; Systolic arterial pressure
MeSH Terms: conditions — Hypovolemia; Coronary Artery Disease; Edema | interventions — Fluid Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fluid Therapy: Systematisation of fluids during CABG surgery
  Interventions: Procedure: Fluids

INTERVENTIONS:
Procedure: Fluids

SUMMARY:
The purpose of this study is to determine if extra systoles can be used to predict fluid responsiveness perioperatively in patients undergoing on pump coronary artery bypass graft (CABG) surgery. As an additional study we will investigate the ability of a mini fluid challenge to predict response of a larger volume of fluid.

DETAILED DESCRIPTION:
From induction of anaesthesia to cardioplegia we will serve two fluid challenges. Before and after each challenge we will collect hemodynamic data and use this to asses our two hypotheses.

Fluid responsiveness (the outcome to predict) will be defined as a 15% increase in stroke volume(SV) from immediately before fluid infusion is initiated (baseline) to after the full fluid infusion. Stroke volume is derived from the gold-standard pulmonary artery catheter measurement of cardiac output(CO), which is standard monitoring for these patients (SV = CO/heart rate). From subsequent offline analysis of the extracted curve data we will investigate if post-ectopic characteristics from identified extra systoles during the baseline period can predict fluid responsiveness (i.e. the SV change). This analysis addresses the primary hypothesis. Also, we will analyse the arterial waveform related to the mini fluid challenge for morphologic changes (comparing heart beats before the infusion with heart beats during the infusion) and see if such transient changes, e.g. in systolic blood pressure, are able to predict fluid responsiveness. This analysis addresses the secondary hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Predominant sinus rhythm (No atrial fibrillation, trigemini, 2nd and 3rd degree atrioventricular block also if pacing is present etc.)

Exclusion Criteria:

* Ejection fraction < 35% (Safety limit minimising risk of fluid overload)
* Haemodialysis (safety precaution for patients with end-stage kidney failure)
* Pregnancy
* Mentally retarded (due to lack of capability to sign an informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for elective on pump CABG surgery at Aarhus University Hospital, SKS.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Cardiac output changes | At 5 minutes
  From initiation of fluid infusion
Systolic arterial pressure changes | 10 minutes prior to fluid infusion
  In relation to extra systoles

SECONDARY OUTCOMES:
Arterial waveform changes | 10 seconds
  From initiation of the mini fluid challenge (part of the compiled fluid challenge)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia and Intensive Care Medicine, Cardiothoracic Anesthesia, Head & Heart Centre, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
No consent for sharing personal data.

REFERENCES:
- [Derived] Berg JM, Nielsen DV, Abromaitiene V, Hjornet NE, Vistisen ST. Changes in arterial blood pressure characteristics following an extrasystolic beat or a fast 50 ml fluid challenge do not predict fluid responsiveness during cardiac surgery. J Clin Monit Comput. 2022 Jun;36(3):889-900. doi: 10.1007/s10877-021-00722-z. Epub 2021 May 26. PMID 34041648